# Official title: Randomized Controlled Trial of a Risk Reframing Tool to Change Mothers' Parenting Associated With Children's Risky Play

NCT number: 03374683

Document date: December 5, 2018

Document type: Informed Consent Form





# Cover Letter Go Play Outside!

## **Title of Project:**

Go Play Outside! Reframing risk to promote children's outdoor play

#### **Principal Investigator**

**Dr. Mariana Brussoni**, Department of Pediatrics, University of British Columbia; BC Children's Hospital.

Email: <a href="mailto:mbrussoni@bcchr.ca">mbrussoni@bcchr.ca</a>; Tel: 604-875-3712

## **Co-Investigators**

**Dr. Louise Masse**, School of Population and Public Health, University of British Columbia; BC Children's Hospital.

Email: <a href="mailto:lmasse@bcchr.ca">lmasse@bcchr.ca</a>; Tel: 604-875-2000 (ext. 5563)

**Dr. Ian Pike**, Department of Pediatrics, University of British Columbia; BC Children's Hospital.

Email: <a href="mailto:ipike@bcchr.ca">ipike@bcchr.ca</a>; Tel: 604-875-3425

#### **Sponsor**

This study is funded by the Lawson Foundation.

## **Purpose**

Outdoor play is important for children as it can promote healthy social and physical development, emotional wellbeing, self-confidence, risk management and overall physical activity. However, opportunities for outdoor play have been decreasing across generations due to perceptions that it is dangerous and unnecessary.

The overarching aim of the Go Play Outside! study is to develop an educational tool to inform parents about the importance of outdoor play for children, and to help them develop strategies for letting children engage in healthy outdoor play.

We are currently conducting Phase 2 of the study where we compare three different educational tools and evaluate how effective each one is, with respect to the others. You are being invited to take part in this study because you are a mother of a child aged between 6 and 12 years, residing in Metro Vancouver area, and can speak, read and understand English.

#### **Study Procedures**

Phase 2 of the Go Play Outside! study will include about 500 mothers of children between the ages of 6 and 12 years, residing in Metro Vancouver. If you agree to participate, you will be asked to complete an online survey and then randomly assigned to one of the three groups: (1) Online Educational Material A group, (2) Online Educational Material B group, or (3) In-Person Workshop group. Neither the researchers, nor you will know in advance which group you will be assigned to. All groups will receive information on the benefits of outdoor play; the difference between the groups is the format, style, and method of delivering the information. If you are assigned to In-Person Workshop group, you will receive an email from us to schedule a time and place for the in-person workshop. There is a 1/3 chance that you are assigned to any group.

Each survey takes about 20 to 30 minutes to complete and you will be invited to take our survey over three time points (i.e., initial time, 1 week after and 3 months after completing the online material or attending the in-person workshop). The total time you will be dedicating to this study will be 45 to 70 minutes if you are assigned to group 1 or 2, or 135 minutes if you are assigned to the in-person workshop.

#### **Potential Risks**

No risks are expected as a result of participating in this study. Nonetheless, if you feel any distress during the study, you can withdraw at any time without any penalty.

#### **Potential Benefits**

While there may not be any direct benefit from participating in this study, potential benefits can result from learning about children's outdoor play, being able to "voice" your opinion and knowing that you are contributing to developing an innovative online tool that educate parents and others about the importance of outdoor play for children.

#### Confidentiality

Your confidentiality will be respected. You will be assigned a unique study number as a participant in this study. This number will not include any personal information that could identify you. Research records and data that can indirectly identifying you (e.g., email address, demographic questions) may, nonetheless, be inspected in the presence of the Principal Investigator by representatives of the Lawson Foundation, Health Canada, and University of British Columbia Research Ethics Board for the purpose of monitoring the research. No information or records that disclose your identity will be published without your consent, nor will any information or records that disclose your identity be removed or released without your consent unless required by law.

Your rights to privacy are legally protected by federal and provincial laws that require safeguards to ensure that your privacy is respected. You also have the legal right of access to the information about you that has been collected for this study, and an opportunity to correct any errors in this information, if needed. Further details about these laws are available on request to your study researcher.

Your survey responses will be stored in a password protected folder in a secured network at the BC Children's Hospital Research for 5 years. Only research staff associated with the project will have access to them for the purpose of data cleaning and analysis. After 5 years, these will be destroyed (i.e., permanently deleted). Any identifiable information (e.g., demographic information, email address) will be encrypted and stored in a password protected folder in a secured network at the BC Children's Hospital or in a locked cabinet at Dr. Brussoni's BC Children's Hospital Research office.

#### **Remuneration/Compensation**

To acknowledge your time and contribution to the study, you will receive \$30 upon completion of the first round of the survey and then \$15 for each follow-up survey you complete (1 week after and 3 months after). For those who are assigned to the In-Person group will receive additional \$30 when attending in-person workshop.

#### Contact for information about the study

If you have any questions or concerns about what we are asking of you, please contact Dr. Mariana Brussoni at <a href="mailto:mbrussoni@bcchr.ca">mbrussoni@bcchr.ca</a> or 604-875-3712; Christina Han, research coordinator at <a href="mailto:chan@bcchr.ca">chan@bcchr.ca</a> or 604-875-2000 ext 2433; or Takuro Ishikawa, graduate academic assistant at <a href="mailto:tishikawa@bcchr.ca">tishikawa@bcchr.ca</a> or 604-875-2000 ext 6708.

## Contact for concerns about the rights of research subjects

If you have any concerns or complaints about your rights as a research participant and/or your experiences while participating in this study, contact the Research Participant Complaint Line in the UBC Office of Research Ethics at 604-822-8598 or if long distance e-mail RSIL@ors.ubc.ca or call toll free 1-877-822-8598.

By completing the survey questionnaire, you are consenting to participate in this research.